CLINICAL TRIAL: NCT07120243
Title: Clinical Effectiveness of Bioactive Silica Based With Calcium Toothpaste, Sodium Fluoride Varnish in Management of White Spot Lesions (A 6m Randomized Clinical Trial).
Brief Title: Clinical Effectiveness of Bioactive Silica Based With Calcium Toothpaste
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rawda Hesham Abd ElAziz (Other)
Responsible Party: Sponsor-Investigator, Rawda Hesham Abd ElAziz, Associate Professor, Conservative dentistry department, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CONS1R
Record Dates: First submitted 2025-06-19; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Caries; Initial; Caries Active
Keywords: Bioactive Silica Based with calcium booster (Refix technology) toothpaste; Caries Prevention; white spot carious lesions
MeSH Terms: interventions — Fluorides, Topical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 Refix Booster: Bioactive Silica Based (Refix technology) with calcium booster toothpaste (Experimental): The patients will be taught in the intervention visit and instructed to use the same 1 inch amount of the two toothpastes, mix them and apply it on a soft bristle toothbrushes with the same brushing technique they for 2 minutes twice a day (morning and last thing at night) along the study period without further rinsing, only spitting of the excess material.
  Interventions: Procedure: Toothpaste Product
- Group 2 Polimo: 5% Sodium Fluoride varnish (Experimental): The tooth will be dried, and cotton roll isolated. According to manufacturer instructions, thin coat of the varnish will be applied on the teeth for 10 - 20 s using a microbrush in a horizontal sweeping motion , then drying with air will be done. Patients will be instructed to avoid food and liquid intake for two hours after varnish application also, to use conventional 1425 ppm fluoride toothpaste at home with the same instructions mentioned before.
  Interventions: Procedure: Varnishes, Fluoride
- Group (3) Signal Complete 8 ; Conventional 1425 ppm fluoride toothpaste: (Active Comparator): The patients will be taught in the intervention visit and instructed to use the same 1 inch amount of the toothpaste and soft bristle toothbrushes with the same brushing technique they for 2 minutes twice a day (morning and last thing at night) along the study period without further rinsing, only spitting of the excess material.
  Interventions: Procedure: Toothpaste Product

INTERVENTIONS:
Procedure: Toothpaste Product — Administration ofa toothpaste
  Arms: Group (3) Signal Complete 8 ; Conventional 1425 ppm fluoride toothpaste:; Group 1 Refix Booster: Bioactive Silica Based (Refix technology) with calcium booster toothpaste
Procedure: Varnishes, Fluoride — The tooth will be dried, and cotton roll isolated. According to manufacturer instructions, thin coat of the varnish will be applied on the teeth for 10 - 20 s using a microbrush in a horizontal sweeping motion , then drying with air will be done.
  Arms: Group 2 Polimo: 5% Sodium Fluoride varnish

SUMMARY:
This study will be conducted to Clinically evaluate Bioactive Silica Based with calcium booster (Refix technology) toothpaste and Sodium Fluoride varnish versus conventional fluoride toothpastes in management of white spot lesions of adult patients over 6m follow up and evaluating patient perception regarding the treatment provided.

ELIGIBILITY:
Inclusion Criteria:

* Patient with non cavitated carious WSL in at least one upper or lower tooth.
* Teeth with active non cavitated white spot carious lesions on the cervical one third of the facial or lingual surfaces.

Teeth with initial carious lesions with score 1 or 2 according to The International Caries Detection and Assessment System (ICDAS).

• Teeth with Diagnodent values between 14-20 that refers to early enamel caries.

Exclusion Criteria:

Patients with known allergies or adverse reactions to any ingredient of the tested materials.

• Systematic disease and/ or physical disabilities that may affect participation.

• Patients with white spots due to congenital reasons e.g. enamel hypomineralization.

• Pregnant females with frequent vomiting attacks.

• Smokers.

• Excessive dietary or environmental exposure to acids.

* Presence of surface cavitation or restorations .

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Degree of Remineralization efficacy by Diagnodent | change from the baseline, 1month, 3 months , 6 months after treatment
  DIAGNOdent calibration will be performed first then the tip of the probe will be positioned on the lesion and rotated around its vertical axis until the highest value will be reached and a peak reading will be recorded

SECONDARY OUTCOMES:
Carie Progression according to International Caries Detection and Assessment System (ICDAS) scale: | change from the baseline, 1month, 3 months , 6 months after treatment
  The tooth will be visually examined according to the ICDAS scale as follows: "Code 0: Sound tooth surface: There should be no evidence of caries.
  Code 1: First visual change in enamel: When seen wet there is no evidence of any change in color attributable to carious activity, but after prolonged air drying a carious opacity (white or brown lesion) is visible that is not consistent with the clinical appearance of sound enamel.
  Code 2: Distinct visual change in enamel when viewed wet: There is a carious opacity or discoloration (white or brown lesion) that is not consistent with the clinical appearance of sound enamel. This lesion may be seen directly when viewed from the buccal or lingual direction. In addition, when viewed from the occlusal direction, this opacity or discoloration may be seen as a shadow confined to enamel, seen through the marginal ridge.
  Code 3: Initial breakdown in enamel due to caries with no visible dentin: Once dried for approximately five seconds there is disti
Patient-reported outcome measures (PROMs): Patients perception of the treatment | change from the baseline, 1month, 3 months , 6 months after treatment
  Patients will be evaluated regarding their perception of the treatment provided outcome using Global Impression of Change Questionnaire (GICQ) which is a seven-point scale describing the overall impression of the patients toward the treatment of the lesions and change from the baseline as follows: 'very much worse', 'worse', 'a little worse', 'unchanged', 'a little better', 'better', 'very much better'. satisfied".

IPD SHARING:
Plan to Share IPD: No